CLINICAL TRIAL: NCT05615298
Title: Multi-reader, Multi-case, Observer-blind, Retrospective, Pivotal Study to Evaluate Effectiveness of Investigational Device in the Assistance of Detection and Diagnosis of Breast Cancer During Screening Mammography Interpretation
Brief Title: Study to Evaluate Effectiveness of Investigational Device in the Assistance of Detection and Diagnosis of Breast Cancer
Status: Completed | Type: Observational
Sponsor: Lunit Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: LUN_MMG_121
Record Dates: First submitted 2022-11-02; First posted 2022-11-14 (Actual); Last update posted 2022-11-14 (Actual); Status verified 2022-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Cancer: * Negative image data: Has been interpreted as negative in screening mammograms
  * Benign image data: Has a suspicious lesion for breast cancer in screening mammograms but confirmed as a benign through the follow-up biopsy or has been interpreted as a benign in screening mammograms and confirmed as a benign in the further diagnostic images taken after at least two years from the screening mammograms.
  Interventions: Radiation: Mammography
- Non-cancer: Has a suspicious lesion for breast cancer in screening mammograms and confirmed as a cancer (malignant) through the follow-up biopsy.
  Interventions: Radiation: Mammography

INTERVENTIONS:
Radiation: Mammography — FFDM (Full-Field Digital mammography)

SUMMARY:
This study aims to evaluate Effectiveness of Investigational Device, Lunit INSIGHT MMG, in the assistance of Detection and Diagnosis of Breast Cancer during Screening Mammography Interpretation.

DETAILED DESCRIPTION:
The Lunit INSIGHT MMG is developed as a computer-assisted detection/diagnosis device based on deep learning technology. In this pivotal study, effectiveness of the investigational device, Lunit INSIGHT MMG, was examined by comparing the reading panelist's interpretation ability between CAD assisted and unassisted during screening mammography interpretation.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Any ethnic origin
* Acquired with devices from two manufacturers: Hologic and GE
* 4 views (RMLO, LMLO, RCC, LCC) images of FFDM (Full-Field Digital mammography)

Exclusion Criteria:

* Previous core needle biopsy in breast for past 2 years
* Previous vacuum-assisted biopsy, surgical biopsy or surgery in breast
* Previous breast cancer
* Lactating when taking screening mammograms
* Presence of a breast implant in screening mammograms
* Presence of a pacemaker in screening mammograms
* Inadequate quality status such as insufficient anatomical coverage of screening mammograms

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Screenign Mammography Population
Sampling Method: Probability Sample
Enrollment: 240 (Actual)
Dates: Start 2020-06-15 (Actual); Primary Completion 2021-01-13 (Actual); Study Completion 2021-01-13 (Actual)

PRIMARY OUTCOMES:
Patient-level FBR (forced BI-RADS) area under the Receiver Operating Characteristic (ROC) curve | Through study completion, an average of 6 months
  Patient-level FBR (forced BI-RADS) area under the Receiver Operating Characteristic (ROC) curve to measure the effectiveness of Investigational Device between CAD assited and unassisted environment

CONTACTS AND LOCATIONS:
Overall Officials: Gregg Miller, MD, Principal Investigator — Atrius Health
Locations (1):
- Atrius Health, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No